CLINICAL TRIAL: NCT04185675
Title: Comparison of Two Types of Videolaryngoscope and Direct Laryngoscope in Expected Non-difficult Airway Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E2019012
Record Dates: First submitted 2019-11-30; First posted 2019-12-04 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Laryngoscopes
Keywords: Visual laryngoscope; Direct laryngoscope; Tracheal intubation time

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Macintosh laryngoscope (Active Comparator)
  Interventions: Device: The laryngoscope used for tracheal intubation under general anesthesia for patients with expected non-difficult airway conditions.
- nonadjustable videolaryngoscope (Experimental)
  Interventions: Device: The laryngoscope used for tracheal intubation under general anesthesia for patients with expected non-difficult airway conditions.
- adjustable videolaryngoscope (Experimental)
  Interventions: Device: The laryngoscope used for tracheal intubation under general anesthesia for patients with expected non-difficult airway conditions.

INTERVENTIONS:
Device: The laryngoscope used for tracheal intubation under general anesthesia for patients with expected non-difficult airway conditions. — All the patients will receive the same anesthesia induction, and are randomized to three groups to receive different types of laryngoscope for intubation. These are the direct Macintosh laryngoscope, adjustable videolaryngoscope and nonadjustable videolaryngoscope.

SUMMARY:
Macintosh direct laryngoscope has been mostly widely used for anesthesiologists in operation rooms or emergency situations all over the world. With rapidly development of technical devices, nowadays videolaryngoscope has become more and more popular in hospitals, for it could improve first intubation success rate and it is easier for beginners to learn. And there are many different types of videolaryngoscope for different purpose, like with or without a channel, different curvature, and so go. In this study, our aim is to study whether the videolaryngoscope which can be adjustable or not costs less intubation time and causes fewer injury in expected non-difficult airway patients by experienced anesthesiologists, compared with the classic Macintosh direct laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* age between18 and 65 years
* ASA(American Society of anesthesiologists) I-II
* BMI 18-30 kg/m2
* scheduled to receive elective surgery under general anesthesia with expected non-difficult airway in operation rooms.

Exclusion Criteria:

* expected difficult airway
* allergy to anesthesia induction drugs
* scheduled to receive surgeries affecting vocalisation
* with high reflux aspiration risk
* with acute and chronic cardiac or respiratory failure
* with glucocorticoids medication history
* with mental disorder or transferred to SICU(Surgical Intensive Care Unit) or ICU after surgery who can not cooperate well with others
* refused or have participated in other clinical trials that may have effects on the outcomes of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Tracheal intubation time | time from the removal of the patient's face mask for preoxygenation to confirmation of good tube position based on continuous positive end-tidal carbon dioxide reading (at least three breaths without a significant visual decrease in capnography).
  total time to successful orotracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Sanqing Jin, Doctor, Study Chair — Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Not decided yet. We plan to share the above information from the article has been published to six months after publication.
Access Criteria: Access Criteria has not been decided.